CLINICAL TRIAL: NCT07089667
Title: The Effect of Virtual Reality Exergame on Physical Activity and Fitness in The Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Andi Amirah Shaleha Junaedi, Principal Investigator, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UH24010039
Record Dates: First submitted 2025-07-07; First posted 2025-07-28 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Healthy Elderly
Keywords: Virtual Reality Exergame; Older Adult; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Exergaming; Congresses as Topic

STUDY DESIGN:
Intervention Model Description: The interventional study model in this research employs a parallel design, where participants are randomly assigned into two groups. One group receives the intervention in the form of Virtual Reality Exergame, while the other group serves as a control group receiving conventional aerobic exercise following the Ministry of Health. Both groups proceed simultaneously throughout the study period to compare the effects of the intervention on physical activity and fitness in older adults. This parallel model allows for a direct evaluation of the effectiveness of Virtual Reality Exergame by comparing outcomes between groups at the same time, resulting in more valid and reliable findings. Randomization is used to minimize bias and ensure equivalence between groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: In this study, masking is applied to both the investigators and the outcomes assessors to minimize bias during data collection and analysis. The investigators who analyze the data are blinded to the participants' group assignments to ensure objective interpretation of the results. The outcomes assessors, responsible for evaluating physical activity and fitness, are also blinded to which intervention each participant received, preventing subjective influence on outcome measurement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality exergame (Experimental): The Virtual Reality Exergame intervention involves physical exercise sessions using VR technology - the game Ring Fit Adventure, specifically designed for older adults. Participants begin with 10-minute exercise sessions, increasing by 5 minutes each week until reaching 30 minutes per session. The exercise frequency is three times per week, conducted over a 6-week period. The exercise prescription follows a protocol developed by the researchers. The training includes aerobic movements integrated into interactive games (types of games as specified in the protocol) that stimulate physical activity and motor coordination.
  Interventions: Behavioral: virtual reality exergame
- Conventional-based aerobic exercise (Active Comparator): The control group performs conventional aerobic exercise based on video aerobic exercise of the Ministry of Health (KEMENKES) protocol, with the same duration and frequency, to ensure an equivalent comparison in improving physical activity and fitness among older adults. Participants begin with 10-minute exercise sessions, increasing by 5 minutes each week until reaching 30 minutes per session. The exercise frequency is three times per week, conducted over a 6-week period. The exercise prescription follows a protocol developed by the researchers.
  Interventions: Behavioral: Conventional

INTERVENTIONS:
Behavioral: virtual reality exergame — virtual reality exergame using Nintendo RingFit
  Arms: virtual reality exergame
Behavioral: Conventional — Conventional-based aerobic exercise using video aerobic exercise of the Ministry of Health (KEMENKES) protocol
  Arms: Conventional-based aerobic exercise

SUMMARY:
Virtual Reality exergame is a video games that combine body motion control with physical activity in a safe virtual environment. In the elderly, VR exergames like the Nintendo Switch RingFit Adventure aid rehabilitation, improving physical function, cognition, balance and mental well-being. These games overcome the boredom of traditional exercise with a multisensory and interactive environment that engages the whole body. The general objective of the present research is to evaluate the effectiveness of virtual reality exergames on physical activity and fitness in the elderly.

Design : This study is an experimental study with a randomized controlled trial - double blind design. This experimental study was conducted with blinding, specifically a single blinding where the researcher and data analyst (statistician) did not know the allocation of samples to the intervention and control groups.

DETAILED DESCRIPTION:
Aging is associated with a decline in biological, physiological, and functional capacities, impacting muscle strength, flexibility, balance, and the ability to perform daily activities. This decline adversely affects the quality of life in the elderly, measurable through the concept of healthy adjusted life expectancy (HALE). In Indonesia, the average HALE is 62.25 years, indicating a loss of approximately 8.85 years due to chronic diseases and disabilities.

One effective strategy to address chronic diseases and disabilities is the implementation of physical activities or exercises, including aerobic, strength, flexibility, and balance training, as recommended by the World Health Organization (WHO). Aerobic exercise not only enhances cardiovascular and pulmonary function but also provides broader benefits to both physical and mental health. However, adherence and motivation in elderly populations are often low due to external factors such as limited mobility and unsupportive environments.

To overcome these challenges, exergames have emerged as an innovative intervention combining active video gaming with physical exercise. Virtual Reality (VR) exergames, such as the Nintendo Switch RingFit Adventure, offer immersive, multisensory, and interactive environments that enhance motivation for exercise among older adults. Evidence suggests that VR exergame interventions can improve physical function, reduce symptoms of depression and anxiety, and enhance health-related quality of life, although research on fitness outcomes in the elderly remains limited and warrants further investigation.

The general objective : to evaluate the effectiveness of virtual reality exergames on physical activity and fitness in the elderly.

Specific objectives:

* To determine the difference in effectiveness between virtual reality exergame and aerobic exercise training on physical activity in the older adult.
* To determine the difference in effectiveness between virtual reality exergame and aerobic exercise training on body composition parameters in the older adult.
* To determine the difference in effectiveness between virtual reality exergame and aerobic exercise training on hand muscle strength parameters in the older adult.
* To determine the difference in effectiveness between virtual reality exergame and aerobic exercise training on muscle endurance in the older adult.
* To determine the difference in effectiveness between virtual reality exergame and aerobic exercise training on flexibility in the older adult.

Methods : This study is an experimental study with a randomized controlled trial - double blind design. The study sample consisted of 40 patients assigned to the intervention group (n=20) or control group (n=20). The study will be conducted from February 2024 to June 2024, targeting the elderly population in Makassar City, South Sulawesi, Indonesia. The accessible population consists of elderly individuals in the Zaitun Elderly Community.

Researcher will compare the intervention group, which participates in virtual reality exergame-based aerobic exercise, with the control group, which engages in video-based aerobic exercise provided by the Ministry of Health, focusing on physical activity and physical fitness outcomes.

* Participants will undergo interviews, physical examinations (vital signs, nutritional status, weight, height, and BMI), and additional assessments before and after 6 weeks of exercise, including :

  1. IPAQ (International Physical Activity Questionnaire) for daily activity, muscle endurance (30-second sit-to-stand test), hand strength (dynamometer), flexibility (chair-sit-and-reach test), and body composition (bioimpedance analysis).
  2. Cognitive function (MOCA-Ina), exercise intensity (Borg Scale), and pre-exercise protocols (risk screening, 6-minute walking test) on the first day, followed by an introduction to equipment and exercise clothing.
* Both groups will follow a warm-up and cool-down routine for 10 minutes before and after exercise. The treatment group will perform VR exergame exercises using Nintendo Switch Ring Fit Adventure 3 times per week for 6 weeks, while the control group will perform conventional aerobic exercises supervised by a doctor.
* Exercise adherence and intensity will be monitored and recorded in a logbook, along with any complaints before, during, and after each session. The estimated time required for each meeting (training session) will increase every week by 40 - 60 minutes.
* At the end of the study, data will be collected again, and any adverse event (AE) experienced by participants will be addressed. Researcher will pause exercises and treat them if symptoms such as cybersickness occur.

Ethical Approval and Sample Criteria This study has obtained ethical approval from the Ethics Committee of the Faculty of Medicine, Hasanuddin University, Makassar, Indonesia, to ensure the quality and compliance of the research.

The data collected will undergo descriptive analysis to outline the characteristics of the participants. For hypothesis testing, chi-square or McNemar tests will be used for categorical dependent variables, while t-tests will analyze numerical dependent variables. The effects of VR exergame compared to aerobic exercise will be assessed using independent t-tests for normally distributed data and Mann-Whitney tests for non-normal data. Normality and homogeneity of numerical dependent variables will be evaluated using the Kolmogorov-Smirnov test, with p-values greater than 0.05 indicating normal distribution. Results will be comprehensively discussed by the research team and experts to draw appropriate conclusions. Correlation between variables will be measured using Pearson's correlation for normally distributed numerical data, Spearman's test for ordinal categorical data, or contingency coefficients for nominal categorical data. All analyses will be conducted using SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study
2. Aged above 60 years
3. Able to watch television with or without glasses from a distance of 2 meters (visual acuity between 20/20 and 20/80)
4. No cognitive impairment (MOCA-Ina score: 26-30)

Exclusion Criteria:

1. Congestive heart failure
2. Uncontrolled hypertension
3. History of fracture or surgery within the last 6 months
4. Currently on the waiting list for orthopedic surgery
5. Myocardial infarction or stroke within the last 6 months
6. Dependence on a wheelchair
7. Severe hearing and vision impairments
8. Other neuromusculoskeletal disorders that interfere with the ability to perform exercises (pain with VAS > 4)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
physical activity | Physical activity was assessed at week 0 (before the intervention) and week 6 (after the intervention) to evaluate changes in participants' physical activity levels during the intervention period.
  Physical activity was measured using the Indonesian version of the International Physical Activity Questionnaire (IPAQ) - Short Form.
  The International Physical Activity Questionnaire (IPAQ) score is calculated by assessing the duration and frequency of physical activities across three categories: walking, moderate-intensity, and vigorous-intensity activities. Each category is assigned a standard Metabolic Equivalent of Task (MET) value, namely 3.3 METs for walking, 4.0 METs for moderate activities, and 8.0 METs for vigorous activities. The weekly total MET-minutes are obtained by multiplying the MET value by the minutes per day and the number of days per week for each activity type, then summing these values across all categories. Based on the total MET-minutes per week, physical activity levels are interpreted :
  * Sedentary (<600 MET-minutes/week)
  * Intermediate (600-3,000 MET-minutes/week)
  * Active (>3,000 MET-minutes/week)
body composition (muscle mass) | Body composition (muscle mass) was assessed at week 0 (before the intervention) and week 6 (after the intervention) to evaluate changes in participants' body composition during the intervention period.
  The body composition (muscle mass) parameter is integratedly measured using Bioelectrical Impedance Analysis (BIA) with the Tanita BC 730 device.
  interpretation : Muscle mass, also presented as a percentage, reflects lean body mass important for function, with males aged 60-79 years ranging from 70-84% and females from 60-72.5%.
Hand muscle strength | Hand muscle strength was assessed at week 0 (before the intervention) and week 6 (after the intervention) to evaluate changes in participants' hand muscle strength during the intervention period.
  Hand muscle strength was measured using an electronic hand dynamometer, CAMRY ISO 9001 model EH101.
Muscle endurance | Muscle endurance was assessed at week 0 (prior to the intervention) and week 6 (post-intervention) to evaluate changes in participants' muscle endurance throughout the intervention period.
  Muscle endurance was measured using the 30-second sit-to-stand test with a stopwatch
Flexibility | Flexibility was assessed at week 0 (prior to the intervention) and week 6 (post-intervention) to evaluate changes in participants' flexibility throughout the intervention period.
  Flexibility was assessed using the Chair Sit-and-Reach Test.
body composition (fat mass) | Body composition (fat mass) was assessed at week 0 (before the intervention) and week 6 (after the intervention) to evaluate changes in participants' body composition during the intervention period.
  The body composition (fat mass) parameter is integratedly measured using Bioelectrical Impedance Analysis (BIA) with the Tanita BC 730 device.
  Interpretation :
  Fat mass is expressed as a percentage of total body weight, varying by age and sex; for instance, males over 40 years typically range from 11-24%, while females range from 23-35%.
Body composition (Bone mass) | Body composition (bone mass) was assessed at week 0 (before the intervention) and week 6 (after the intervention) to evaluate changes in participants' body composition during the intervention period.
  The body composition (bone mass) parameter is integratedly measured using Bioelectrical Impedance Analysis (BIA) with the Tanita BC 730 device.
  interpretation : Bone mass is reported in kilograms and stratified by weight and sex, such as 2.65-3.29 kg for males weighing 65-95 kg and about 2.40 kg for females weighing between 50-75 kg.

CONTACTS AND LOCATIONS:
Overall Officials: Andi Amirah Shaleha Junaedi, MD, M.Sc, Principal Investigator — Physical Medicine and Rehabilitation, Faculty of Medicine of Hasanuddin University, Indonesia
Locations (1):
- GPIB Jemaat Bukit Zaitun, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
we plan to share all collected individual participant data (IPD) as well as all IPD that underlie the results reported in any publications arising from this study. This will ensure transparency and allow other researchers to verify, replicate, or build upon our findings.
Supporting Information: Study Protocol, CSR
Time Frame: The individual participant data (IPD) and accompanying supporting information will be made available starting 6 months after the publication of the main study results and will remain accessible for a period of 5 years. This timeframe allows sufficient time for initial data analysis and dissemination, while providing other researchers ample opportunity for secondary analysis and collaboration.
Access Criteria: Access to individual participant data (IPD) and supporting documentation will be granted to qualified researchers who submit a formal request outlining the purpose and proposed analyses. Data will be shared for purposes consistent with advancing scientific knowledge in the field of physical activity, virtual reality, aging. Requests will be reviewed by the principal investigator and a data access committee to ensure ethical use and participant confidentiality. Data will be shared through a secure data-sharing platform after signing a data use agreement to protect privacy and intellectual property

REFERENCES:
- [Background] Riebe, D. (2018) ACSM's Guidelines for Exercise Testing and Prescription. Tenth, Wolters Kluwer. Tenth. Edited by J.K. Ehrman, G. Liguori, and M. Magal. philadelphia: Wolters Kluwer.
- [Background] Yeom HA, Jung D, Choi M. Adherence to Physical Activity Among Older Adults Using a Geographic Information System: Korean National Health and Nutrition Examinations Survey IV. Asian Nurs Res (Korean Soc Nurs Sci). 2011 Jun;5(2):118-27. doi: 10.1016/S1976-1317(11)60020-0. Epub 2011 Jul 8. PMID 25030261
- [Result] Matos-Duarte M, Martínez-de-Haro V, Sanz-Arribas I, Berlanga LA. Functional flexibility in institutionalized sedentary older adults. Rev Bras Cineantropom Desempenho Hum 2021, 23:e73816. DOI: http://doi.org/10.1590/19800037.2021v23e73816
- [Result] Mologne MS, Hu J, Carrillo E, Gomez D, Yamamoto T, Lu S, Browne JD, Dolezal BA. The Efficacy of an Immersive Virtual Reality Exergame Incorporating an Adaptive Cable Resistance System on Fitness and Cardiometabolic Measures: A 12-Week Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Dec 23;20(1):210. doi: 10.3390/ijerph20010210. PMID 36612530
- [Result] Alcazar J, Alegre LM, Van Roie E, Magalhaes JP, Nielsen BR, Gonzalez-Gross M, Judice PB, Casajus JA, Delecluse C, Sardinha LB, Suetta C, Ara I. Relative sit-to-stand power: aging trajectories, functionally relevant cut-off points, and normative data in a large European cohort. J Cachexia Sarcopenia Muscle. 2021 Aug;12(4):921-932. doi: 10.1002/jcsm.12737. Epub 2021 Jul 3. PMID 34216098
- [Result] Munoz-Bermejo L, Adsuar JC, Mendoza-Munoz M, Barrios-Fernandez S, Garcia-Gordillo MA, Perez-Gomez J, Carlos-Vivas J. Test-Retest Reliability of Five Times Sit to Stand Test (FTSST) in Adults: A Systematic Review and Meta-Analysis. Biology (Basel). 2021 Jun 9;10(6):510. doi: 10.3390/biology10060510. PMID 34207604
- [Result] Feodoroff B, Konstantinidis I, Frobose I. Effects of Full Body Exergaming in Virtual Reality on Cardiovascular and Muscular Parameters: Cross-Sectional Experiment. JMIR Serious Games. 2019 Aug 28;7(3):e12324. doi: 10.2196/12324. PMID 31464194
- [Result] Jin, M.. (2023). EFFECTS OF AEROBIC EXERCISE ON BODY MORPHOLOGY IN OBESE UNIVERSITY STUDENTS. Revista Brasileira De Medicina Do Esporte, 29, e2022_0221. https://doi.org/10.1590/1517-8692202329012022_0221
- [Result] Leiros-Rodriguez R, Soto-Rodriguez A, Perez-Ribao I, Garcia-Soidan JL. Comparisons of the Health Benefits of Strength Training, Aqua-Fitness, and Aerobic Exercise for the Elderly. Rehabil Res Pract. 2018 Jun 19;2018:5230971. doi: 10.1155/2018/5230971. eCollection 2018. PMID 30018825
- [Result] Nishi, N. , Tanaka, N. and Hirano, N. (2022) Characteristics of Body Composition and Relationship between Muscle Mass and Muscle Strength among Elderly Women in Different Age Groups. Advances in Aging Research, 11, 135-149. doi: 10.4236/aar.2022.115010.
- [Result] Bai X, Soh KG, Omar Dev RD, Talib O, Xiao W, Soh KL, Ong SL, Zhao C, Galeru O, Casaru C. Aerobic Exercise Combination Intervention to Improve Physical Performance Among the Elderly: A Systematic Review. Front Physiol. 2022 Jan 4;12:798068. doi: 10.3389/fphys.2021.798068. eCollection 2021. PMID 35058805
- [Result] Rodriguez-Almagro D, Achalandabaso-Ochoa A, Ibanez-Vera AJ, Gongora-Rodriguez J, Rodriguez-Huguet M. Effectiveness of Virtual Reality Therapy on Balance and Gait in the Elderly: A Systematic Review. Healthcare (Basel). 2024 Jan 9;12(2):158. doi: 10.3390/healthcare12020158. PMID 38255047
- [Result] Naugle KE, Cervantes XA, Boone CL, Wind B, Naugle KM. Exploring actual and perceived levels of physical activity intensity during virtual reality active games. Front Sports Act Living. 2024 Feb 9;6:1349521. doi: 10.3389/fspor.2024.1349521. eCollection 2024. PMID 38406766
- [Result] Janeh O, Frundt O, Schonwald B, Gulberti A, Buhmann C, Gerloff C, Steinicke F, Potter-Nerger M. Gait Training in Virtual Reality: Short-Term Effects of Different Virtual Manipulation Techniques in Parkinson's Disease. Cells. 2019 May 6;8(5):419. doi: 10.3390/cells8050419. PMID 31064145
- [Result] Dore B, Gaudreault A, Everard G, Ayena JC, Abboud A, Robitaille N, Batcho CS. Acceptability, Feasibility, and Effectiveness of Immersive Virtual Technologies to Promote Exercise in Older Adults: A Systematic Review and Meta-Analysis. Sensors (Basel). 2023 Feb 24;23(5):2506. doi: 10.3390/s23052506. PMID 36904709
- [Result] Gao Z, Lee JE, McDonough DJ, Albers C. Virtual Reality Exercise as a Coping Strategy for Health and Wellness Promotion in Older Adults during the COVID-19 Pandemic. J Clin Med. 2020 Jun 25;9(6):1986. doi: 10.3390/jcm9061986. PMID 32630367
- [Result] Campo-Prieto P, Cancela-Carral JM, Rodriguez-Fuentes G. Feasibility and Effects of an Immersive Virtual Reality Exergame Program on Physical Functions in Institutionalized Older Adults: A Randomized Clinical Trial. Sensors (Basel). 2022 Sep 6;22(18):6742. doi: 10.3390/s22186742. PMID 36146092
- [Result] Kruse, L., Karaosmanoglu, S., Rings, S., Ellinger, B., & Steinicke, F. (2021). Enabling Immersive Exercise Activities for Older Adults: A Comparison of Virtual Reality Exergames and Traditional Video Exercises. Societies, 11(4), 134. https://doi.org/10.3390/soc11040134
- [Result] Triangto K, Radi B, Siswanto BB, Tambunan TF, Heriansyah T, Harahap AR, Kekalih A, Katsukawa H, Santoso A. Non-dominant handgrip strength is associated with higher cardiorespiratory endurance and elevated NT-proBNP concentrations in ambulatory male adult outpatients with stable HFrEF. Narra J. 2024 Dec;4(3):e1278. doi: 10.52225/narra.v4i3.1278. Epub 2024 Nov 25. PMID 39816091
- [Result] Li M, Ogilvie H, Ochala J, Artemenko K, Iwamoto H, Yagi N, Bergquist J, Larsson L. Aberrant post-translational modifications compromise human myosin motor function in old age. Aging Cell. 2015 Apr;14(2):228-35. doi: 10.1111/acel.12307. Epub 2015 Feb 2. PMID 25645586
- [Result] Yang CM, Chen Hsieh JS, Chen YC, Yang SY, Lin HK. Effects of Kinect exergames on balance training among community older adults: A randomized controlled trial. Medicine (Baltimore). 2020 Jul 10;99(28):e21228. doi: 10.1097/MD.0000000000021228. PMID 32664177
- [Result] Tuan SH, Chang LH, Sun SF, Lin KL, Tsai YJ. Using exergame-based exercise to prevent and postpone the loss of muscle mass, muscle strength, cognition, and functional performance among elders in rural long-term care facilities: A protocol for a randomized controlled trial. Front Med (Lausanne). 2022 Dec 13;9:1071409. doi: 10.3389/fmed.2022.1071409. eCollection 2022. PMID 36582297
- [Result] Brady, N., McVeigh, J. G., McCreesh, K., Rio, E., Dekkers, T., & Lewis, J. S. (2021). Exploring the effectiveness of immersive Virtual Reality interventions in the management of musculoskeletal pain: a state-of-the-art review. Physical Therapy Reviews, 26(4), 262-275. https://doi.org/10.1080/10833196.2021.1903209
- [Result] Maddison R, Foley L, Ni Mhurchu C, Jiang Y, Jull A, Prapavessis H, Hohepa M, Rodgers A. Effects of active video games on body composition: a randomized controlled trial. Am J Clin Nutr. 2011 Jul;94(1):156-63. doi: 10.3945/ajcn.110.009142. Epub 2011 May 11. PMID 21562081
- [Result] Karahan AY, Tok F, Taskin H, Kucuksarac S, Basaran A, Yildirim P. Effects of Exergames on Balance, Functional Mobility, and Quality of Life of Geriatrics Versus Home Exercise Programme: Randomized Controlled Study. Cent Eur J Public Health. 2015 Nov;23 Suppl:S14-8. doi: 10.21101/cejph.a4081. PMID 26849537
- [Result] Maillot P, Perrot A, Hartley A. Effects of interactive physical-activity video-game training on physical and cognitive function in older adults. Psychol Aging. 2012 Sep;27(3):589-600. doi: 10.1037/a0026268. Epub 2011 Nov 28. PMID 22122605
- [Result] Fragala MS, Cadore EL, Dorgo S, Izquierdo M, Kraemer WJ, Peterson MD, Ryan ED. Resistance Training for Older Adults: Position Statement From the National Strength and Conditioning Association. J Strength Cond Res. 2019 Aug;33(8):2019-2052. doi: 10.1519/JSC.0000000000003230. PMID 31343601
- [Result] Shahana, A., Nair, U.S. and Hasrani, S.S. (2010) 'Effect of aerobic exercise programme on health related physical fitness components of middle aged women', British Journal of Sports Medicine, 44(Suppl_1), pp. i19-i19. Available at: https://doi.org/10.1136/bjsm.2010.078725.60.
- [Result] Haley C, Andel R. Correlates of physical activity participation in community-dwelling older adults. J Aging Phys Act. 2010 Oct;18(4):375-89. doi: 10.1123/japa.18.4.375. PMID 20956840
- [Result] Lo YP, Chiang SL, Lin CH, Liu HC, Chiang LC. Effects of Individualized Aerobic Exercise Training on Physical Activity and Health-Related Physical Fitness among Middle-Aged and Older Adults with Multimorbidity: A Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Dec 25;18(1):101. doi: 10.3390/ijerph18010101. PMID 33375668
- See also: Effects of Individualized Aerobic Exercise Training on Physical Activity and Health-Related Physical Fitness among Middle-Aged and Older Adults with Multimorbidity: A Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/33375668/
- See also: WHO - Multisectoral action for a life course approach to healthy ageing: draft global strategy and plan of action on ageing and health — https://apps.who.int/gb/ebwha/pdf_files/WHA69/A69_17-en.pdf
- See also: WHO guidelines on physical activity and sedentary behaviour — https://www.who.int/publications/i/item/9789240015128
- See also: EFFECT OF AEROBIC EXERCISE ON PHYSICAL FUNCTION INDICES IN THE ELDERLY — https://www.scielo.br/j/rbme/a/sJJLhnrNn5G8FymrgdK46CC/#
- See also: The effect of low impact aerobic exercise on increasing physical fitness for the elderly — https://scholarhub.uny.ac.id/cgi/viewcontent.cgi?article=1034&context=jolahraga
- See also: EFFECT OF AEROBIC EXERCISE ON NEUROMUSCULAR QUALITY IN THE ELDERLY — https://www.scielo.br/j/rbme/a/Gy99C9ycgYZkh8wLLyrFxFP/
- See also: Effects of virtual reality-based aerobic endurance training on the functional fitness of healthy older adults: A systematic review — https://www.researchgate.net/publication/360905190_Effects_of_virtual_reality-based_aerobic_endurance_training_on_the_functional_fitness_of_healthy_older_adults_A_systematic_review
- See also: The Effect Of Aerobic Exercise On Body Weight and Body Fat Percentage — https://eudl.eu/doi/10.4108/eai.28-4-2021.2312189
- See also: EFFECT OF AEROBIC EXERCISE ASSOCIATED WITH RESISTANCE TRAINING ON BODY COMPOSITION OF MIDDLE-AGED AND ELDERLY WOMEN — https://www.scielo.br/j/rbme/a/ypmRHWPjjT5f8dT77CwqKns/?format=pdf&lang=en
- Available data/document: Study Protocol — https://drive.google.com/drive/folders/1QpzE6ACGieVNCGQ1nsLJHxUWtB-fUfLV?usp=sharing

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-08-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT07089667/Prot_SAP_ICF_000.pdf